CLINICAL TRIAL: NCT03200613
Title: Apixaban Versus Low-Molecular Weight Heparin For Thromboprophylaxis In Patients With Acute Spinal Cord Injury: A Pilot Study
Brief Title: Apixaban For Thromboprophylaxis In Patients With Acute Spinal Cord Injury
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study not feasible due to too slow recruitment
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Sam Schulman, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SCI Pilot RCT
Record Dates: First submitted 2017-06-21; First posted 2017-06-27 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Spinal Cord Injuries; Venous Thromboembolism
Keywords: Spinal cord injury; Venous thromboembolism; Hemorrhage
MeSH Terms: conditions — Spinal Cord Injuries; Venous Thromboembolism; Hemorrhage | interventions — apixaban; Heparin, Low-Molecular-Weight; Enoxaparin; Dalteparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apixaban (Experimental): Apixaban 2.5 mg orally twice daily
  Interventions: Drug: Apixaban
- Low Molecular Weight Heparin (Active Comparator): Either enoxaparin 40 mg or dalteparin 5000 units subcutaneously once daily
  Interventions: Drug: Low molecular weight heparin

INTERVENTIONS:
Drug: Apixaban — 2.5 mg orally twice daily
  Other Names: Eliquis
  Arms: Apixaban
Drug: Low molecular weight heparin — Dalteparin 5000 units daily or Enoxaparin 40 mg subcutaneous daily
  Other Names: Lovenox or Fragmin
  Arms: Low Molecular Weight Heparin

SUMMARY:
Thromboprophylaxis options are limited for patients with acute spinal cord injury (SCI) and there are no studies on direct oral anticoagulants (DOACs) for thromboprophylaxis in this population. Participants will be randomized to apixaban 2.5 mg twice daily or standard dose low-molecular-weight heparin (LMWH), either enoxaparin 40 mg or dalteparin 5000 units, subcutaneously once daily for 90 days or until fully mobilized, whatever comes first. Thromboprophylaxis will be started as soon as hemostasis is achieved. The primary outcome for this pilot study will be the recruitment rate per year (i.e. the screened to enrolled ratio). The primary efficacy endpoint will be a composite of symptomatic, objectively verified, venous thromboembolism (VTE), defined as upper or lower limb deep vein thrombosis (DVT) and/or pulmonary embolism (PE) or sudden death where PE cannot be excluded. The primary safety endpoint will be major bleeding.

DETAILED DESCRIPTION:
Patients with acute (SCI) have a high risk of VTE despite thromboprophylaxis. The current standard thrombprophylaxis is to use LMWH fas soon as hemostasis is achieved. The duration of thromboprophylaxis is commonly 3 months. This entails once or twice daily subcutaneous injections of LMWH for the patients for this duration, which is inconvenient for the patients. There are currently no studies on use of DOACs for thromboprophylaxis in patients with SCI.

We will perform a pilot study at Hamilton General on apixaban versus LMWH for thromboprophylaxis in patients with acute SCI. Upon providing written informed consent, eligible patients will be randomized to apixaban 2.5 mg twice daily or LMWH, either enoxaparin 40 mg or dalteparin 5000 units, subcutaneously once daily for 90 days or until fully mobilized, whatever comes first.

The primary outcome for the feasibility study will be the recruitment rate per year (i.e. the screened to enrolled ratio). Other key feasibility measures will be accrual ratio, protocol violations pertaining to eligibility criteria and randomization procedures, retention rate for primary end-point assessment at 1 year, and the estimates of endpoint rates in the population. The primary efficacy endpoint will be a composite of symptomatic, objectively verified VTE (upper or lower limb DVT and/or PE) or sudden death where PE cannot be excluded. The primary safety endpoint will be major bleeding.

This will be the first study comparing the use of LMWH against a DOAC in SCI patients. Use of a DOAC such as apixaban can eliminate the burden associated with daily injections for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) with acute spinal cord injury (SCI) presenting to the hospital within 1 week of SCI and is at least 36 h after the injury
* Traumatic SCI
* SCI with or without other injuries

Exclusion Criteria:

* Already on therapeutic oral anticoagulation prior to enrollment
* Active bleeding, intracranial or perispinal hematoma, or acquired or congenital bleeding disorder
* Pregnancy or breast feeding
* Severe renal failure (creatinine clearance ≤30 ml/min)
* Liver cirrhosis
* Severe thrombocytopenia (platelets <50)
* Attending physician believes that the patient is not suitable for the study (for example, psychiatric disorder; history of non-compliance)
* Geographic inaccessibility: planned transfer to other site where follow-up not possible
* Failure to obtain written consent
* Previous hypersensitivity reaction to study drugs
* Patients with expected short hospital admission (≤7 days) due to minor injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Primary feasibility outcome: recruitment rate per year (i.e. the screened to enrolled ratio) | 24 months
  The investigators define success as the ability to identify 20 eligible patients at each center per 12-month period.

SECONDARY OUTCOMES:
Composite of Symptomatic Venous Thromboembolism or Sudden Death Where Pulmonary Embolism Cannot be Excluded | 24 months
  A composite of symptomatic, objectively verified VTE (upper or lower limb DVT and/or PE) or sudden death where PE cannot be excluded
Major Bleeding | 24 months
  Major bleeding according to the International Society on Thrombosis and Haemostasis definition

CONTACTS AND LOCATIONS:
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piran S, Schulman S. Incidence and risk factors for venous thromboembolism in patients with acute spinal cord injury: A retrospective study. Thromb Res. 2016 Nov;147:97-101. doi: 10.1016/j.thromres.2016.09.030. Epub 2016 Oct 3. PMID 27721141
- [Background] Piran S, Schulman S. Thromboprophylaxis in Patients with Acute Spinal Cord Injury: A Narrative Review. Semin Thromb Hemost. 2019 Mar;45(2):150-156. doi: 10.1055/s-0039-1678720. Epub 2019 Feb 11. PMID 30743281